CLINICAL TRIAL: NCT06344377
Title: The Impact of Betaine Supplementation on Body Composition and Lipid Metabolism in a Group of Overweight and Obese Women
Brief Title: Betaine Supplementation and Lipid Metabolism in Overweight and Obese Pre-menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Agata Chmurzyńska, Professor, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BETadiposeWOMEN
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betaine (Experimental): Betaine supplementation for 8 weeks, daily dose of 3 g/d, taken twice a day in a capsulated form. One capsule will contain 500 mg betaine. Daily number of capsules will be 2 x 3 = 6.
  Interventions: Dietary Supplement: Betaine
- Placebo (Placebo Comparator): Placebo will be inactive substance (maltodextrin) provided in the same-looking capsules as betaine. Placebo will be administered twice a day, daily number of capsules will be 2 x 3 = 6.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Betaine — Betaine supplemented for 8 weeks
  Arms: Betaine
Dietary Supplement: Placebo — Placebo supplementation for 8 weeks
  Arms: Placebo

SUMMARY:
Obesity represents a serious global health issue with significant consequences, including an increased risk of chronic diseases. Statistics indicate a growing trend of obesity, highlighting the need to seek methods that improve fat tissue metabolism and reduce obesity-related complications. Previous research on animals has shown that betaine, a substance engaged in one-carbon metabolism, may enhance fat oxidation and lower adipose tissue. Therefore, the aim of the research will be to assess the impact of 8-week betaine supplementation on body composition and lipid metabolism markers, as well as expression of genes related to lipid metabolism, in a group of adult women with abdominal obesity.

This study is designed in a placebo-controlled, double-blinded, randomized fashion. The participants will be overweight or obese pre-menopausal females. Upon enrollment, participants will be randomly assigned to one of two parallel groups: betaine (3g/d) or placebo. The supplementation period will last for 8 weeks. There will be three study meetings: T1 before supplementation, T2 after 4 weeks of supplementation, and T3 after 8 weeks of supplementation. Blood will be drawn and body composition measured, and adipose tissue biopsy taken at meetings T1 and T3. The T2 meeting will involve only body composition measurement. Study outcomes will include body mass and composition (including body fat percent), lipid profile, and the expression of genes related to lipid metabolism in adipose tissue and peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* females
* age: 18-45 years
* pre-menopausal
* overweight or obese: BMI >25 kg/m2
* waist circumference > 80 cm

Exclusion Criteria:

* males
* age <18 or >45 years
* perimenopausal or postmenopausal
* BMI < 25 kg/m2
* waist circumference < 80 cm
* betaine administration for 3 months prior to study
* pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Body composition | 8 weeks, three measurements: at week 0, 4 and 8
  Body composition will include percent body fat and lean body mass measured with air displacement plethysmography
Body mass | 8 weeks, three measurements: at week 0, 4 and 8
  Measured in kg
Waist and hips circumference | 8 weeks, three measurements: at week 0, 4 and 8
  Measured in cm
Lipid profile | 8 weeks, two measurements: at week 0 and 8
  Total cholesterol, Triacylglycerols, LDL-cholesterol, HDL-cholesterol
Gene expression | 8 weeks, two measurements: at week 0 and 8
  Included genes relate to lipid metabolism in adipose tissue: PPARG, CD36, FABP4, UCP1, PPARGC1A, LEP, ADIPOQ, INSR, IRS1, DGAT2, SREBF1, ELOVL5 , FADS3, FASN

SECONDARY OUTCOMES:
Liver function test | 8 weeks, two measurements: at week 0 and 8
  activities of enzymes: ALT, AST, GGTP, ALP
Dietary intake | 8 weeks, two measurements: at week 0 and 8
  Based on food diary
sex hormones | 8 weeks, two measurements: at week 0 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Agata Chumrzynska, Principal Investigator — Poznan University of Life Sciences
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No